CLINICAL TRIAL: NCT06005428
Title: A Phase 2A, Investigator & Subject Blinded, Sponsor Unblinded, Placebo-Controlled, Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics of CRD-4730 in Participants With Catecholaminergic Polymorphic Ventricular Tachycardia
Brief Title: Effectiveness of CRD-4730 in Participants With Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT)
Acronym: CPVT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The early termination of the clinical trial is due to an internal administrative and business decision, the study is not being terminated for safety reasons.
Sponsor: Cardurion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRD-4730-201
Record Dates: First submitted 2023-08-08; First posted 2023-08-22 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: CPVT1; Heart Defects, Congenital; Heart Diseases; Ventricular Tachycardia
Keywords: CaMKII; Catecholaminergic polymorphic VT; Ventricular Tachycardia; CRD-4730
MeSH Terms: conditions — Heart Defects, Congenital; Heart Diseases; Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: 3-period randomized 2-sequence study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator and Subject Blinded, Sponsor Unblinded; Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose 1 (Experimental): CRD-4730 Dose 1 capsule
  Interventions: Drug: CRD-4730
- Dose 2 (Experimental): CRD-4730 Dose 2 capsule
  Interventions: Drug: CRD-4730
- Dose 3 (Placebo Comparator): Placebo capsule to match CRD-4730
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CRD-4730 — Oral CRD-4730 in capsule form
  Arms: Dose 1; Dose 2
Drug: Placebo — Placebo to match CRD-4730 in capsule form
  Arms: Dose 3

SUMMARY:
This is a Phase 2, multicenter, double-blind, sponsor unblinded, placebo-controlled, single-dose clinical study of CRD-4730 to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of CRD-4730 when administered as single oral doses to participants with Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT). The study will have 2 cohorts in which participants with CPVT will participate in a 3-period, randomized 2-sequence study. Each participant will receive 2 different doses of CRD-4730 and 1 dose of matching placebo, with each study drug administered as a single dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females ≥18 years of age, at screening.
2. Confirmed CPVT diagnosis, based on genetic screening for a known RyR2 mutation and a clinical phenotype consistent with CPVT at screening.
3. The participant can perform an EST during which frequent premature ventricular contraction (PVCs) (≥10 per minute), ventricular bigeminy, or higher-grade VA (equivalent to a VA score ≥2) are identified by the investigator.
4. Stable doses of any anti-arrhythmic medication, except amiodarone, for 4 weeks prior to screening.
5. Adhere to all contraceptive criteria.

Exclusion Criteria:

1. Clinically significant structural heart disease, diagnosis of heart failure, or clinically significant coronary artery disease.
2. History of a myocardial infarction, cerebrovascular accident, or transient ischemic attack within 3 months of screening.
3. History of malignancy within the past 5 years at screening (except successfully treated basal cell carcinoma or non-metastatic squamous cell carcinoma of the skin or cervical carcinoma in situ).
4. Female participant that is pregnant or lactating/ breastfeeding, or has plans to do so during the study or within 3 months following last dose of study drug.
5. Use of amiodarone with 3 months prior to screening. NOTE: other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) | Baseline to Day 22
  The number of participants with TEAEs including drug-related AEs, serious AEs (SAEs), and AEs leading to study drug discontinuation will be assessed.
Changes in Laboratory Assessments | Baseline to Day 15
  The number of participants who have normal/ abnormal values at Baseline compared to normal/ abnormal values post-Baseline will be assessed for hematology, serum chemistry and urinalysis.
Changes in Vital Signs Measurement: Systolic and Diastolic blood pressure | Baseline to Day 15
  Percent change from Baseline to post Baseline will be assessed for systolic and diastolic blood pressure
Changes in Vital Signs Measurement: Pulse Rate | Baseline to Day 15
  Percent change from Baseline to post Baseline will be assessed for pulse rate
Changes in Vital Signs Measurement: Respiratory Rate | Baseline to Day 15
  Percent change from Baseline to post Baseline will be assessed for respiratory rate
Changes in Vital Signs Measurement: Body Temperature | Baseline to Day 15
  Percent change from Baseline to post Baseline will be assessed for body temperature
Changes in Physical Exam | Baseline to Day 22
  General physical exams will be carried out to detect any abnormalities in the cardiovascular, respiratory and other body systems
Changes in Electrocardiogram (ECG) Measurements | Baseline to Day 22
  Number of participants who have normal/abnormal ECG measurements at Baseline will be compared to normal/abnormal ECG measurement post Baseline

SECONDARY OUTCOMES:
Change in Ventricular Arrhythmia (VA) score during Exercise Stress Test (EST) | Baseline to Day 1
  The VA score is a physician administered score on a scale of 0-5 with higher numbers being worse.
Change in Ventricular Arrhythmia (VA) score during Exercise Stress Test (EST) | Baseline to Day 8
  The VA score is a physician administered score on a scale of 0-5 with higher numbers being worse.
Change in Ventricular Arrhythmia (VA) score during Exercise Stress Test (EST) | Baseline to Day 15
  The VA score is a physician administered score on a scale of 0-5 with higher numbers being worse.
Assessment of PK effect | Baseline through Day 15
  Plasma concentrations of CRD-4730 over time for each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Jason Homsy, M.D., Ph.D., Study Director — Executive Medical Director
Locations (11):
- United States (3):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Children's Hospital, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas
- Canada (4):
  - Stollery Children's Hospital University of Alberta, Edmonton, Alberta
  - University of British Columbia (UBC) Hospital, Vancouver, British Columbia
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - University of Western Ontario, London, Ontario
- France (3):
  - Hôptal Nord Laennec, Nantes, Loire-Atlantique
  - Hôpital Louis Pradel, Bron
  - Groupe Hospitalier Bichat Claude Bernard, Paris
- IRCCS Pavia Istituti Clinici Scientifici Maugeri Spa Società Benefit, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No